CLINICAL TRIAL: NCT05458596
Title: Nursing Students' Learning About Intimate Partner Violence Against Women With the Screen-based Simulation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gamze Agartioglu Kundakci, PhD(c), Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1212
Record Dates: First submitted 2022-07-08; First posted 2022-07-14 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Nursing Student
Keywords: intimate partner violence; nursing student; screen-based simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screen-based simulation (Experimental): Screen-based simulation about intimate partner violence against women prepared by researchers will apply to nursing students.
  Interventions: Behavioral: Screen-based simulation

INTERVENTIONS:
Behavioral: Screen-based simulation — In the research, training will be given to the sample group on intimate partner violence against women through screen-based simulation.

SUMMARY:
The aim of this research is to develop training material on intimate partner violence against women for nursing students by using the screen-based simulation method.

DETAILED DESCRIPTION:
Intimate partner violence (ipv) against women is characterized as a global epidemic in health care delivery due to its prevalence, high morbidity, and mortality. One of the first healthcare providers that victims interact with is nurses. Nurses should have sufficient knowledge and skills to fulfill their roles and responsibilities defined in the issue of ipv against women. Educational environments must provide nursing students with the opportunity to be aware of ipv against women and to manage cases. Institutions that add simulation content to their education programs have the potential to become the gold standard when preparing nursing students for case management of ipv against women. Screen-based simulations (SBSs) use available digital technology to represent patients, populations, or other healthcare encounters on a computer screen or a mobile tablet, smartphone, or other screen-based devices. Simulations using screens have advantages over mannequin-based simulations-the software is infinitely replicable, the simulation programs can be portable, they can be accessed asynchronously without a live instructor present, and the software can be distributed to many devices, and the programming can track massive amounts of usage data. The aim of this research is to develop training material on intimate partner violence against women for nursing students by using the screen-based simulation method. The sample group of the research in a quasi-experimental design in a single-group pre-test-post-test order will consist of fourth-year students from a university's faculty of nursing. Power analysis was made for the sample size, and it was planned to include 50 students in the sample group. In the research, training will be given to the sample group on ipv against women through screen-based simulation. The research outputs will be measured by Health Workers' Attitudes and Practices on Intimate Partner Violence Against Women Scale, Simulation Design Scale and Debriefing Experience Scale.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being a 4th-year student in the nursing department

Exclusion Criteria:

* Having worked as a nurse before
* To have taken an elective course on violence against women in undergraduate education
* To be married

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The Attitudes and Practices of Healthcare Providers Regarding Intimate Partner Violence (APHCPs-IPV) survey scale | Before the recruit pre-test (APHCPs-IPV survey scale) will be applied. Two weeks after the intervention post-test (APHCPs-IPV survey scale) again will be applied.
  The Turkish version of the scale of 42 items and consists of eight subscales. The subscales are (a) preparedness, (b) self-confidence of the practitioner, (c) lack of control, (d) comfort following disclosure, (e) professional support, (f) practice pressures, (g) abuse inquiries, and (h) practitioner consequences of asking. It is scored on a 4-point scale ranging from 1 to 4 (1- strongly agree, 2 agree, 3-disagree, and 4-strongly disagree). The APHCPs-IPV scale total scores range from 42 to 168. Higher scores reflected greater self-reported preparedness, self-confidence, feelings of professional support, comfort with abuse inquiries, and comfort with discussions following disclosure as well as decreased concern about the consequences of abuse inquiries and decreased feelings of no control and system pressures.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Nursing Faculty, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No